CLINICAL TRIAL: NCT02021838
Title: Evaluation of the Domestic Violence Homicide Prevention Initiative
Brief Title: Evaluation of the Office on Violence Against Women's Domestic Violence Homicide Prevention Demonstrative Initiative
Acronym: DVHPDI
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Sponsor
Other Study IDs: 1311013010
Record Dates: First submitted 2013-12-12; First posted 2013-12-27 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Domestic Violence
Keywords: domestic violence homicide prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- California: Lethality Assessment Program
  Interventions: Other: Lethality Assessment Program
- North Carolina: Lethality Assessment Program
  Interventions: Other: Lethality Assessment Program
- Ohio: Domestic Violence High Risk Team
  Interventions: Other: Domestic Violence High Risk Team
- Illinois: Lethality Assessment Program
  Interventions: Other: Lethality Assessment Program
- Michigan: Lethality Assessment Program
  Interventions: Other: Lethality Assessment Program
- Tennessee: Lethality Assessment Program
  Interventions: Other: Lethality Assessment Program

INTERVENTIONS:
Other: Lethality Assessment Program — Law enforcement officers conduct risk screen of domestic violence victims, if high risk victims are referred to domestic violence services.
  Other Names: LAP
  Groups: California; Illinois; Michigan; North Carolina; Tennessee
Other: Domestic Violence High Risk Team — Law enforcement officers conduct risk screen of domestic violence victims, if high risk victims are referred to domestic violence services and a team who monitors the clinical and criminal justice progress.
  Other Names: HRT
  Groups: Ohio

SUMMARY:
In collaboration with the National Institute of Justice (NIJ) and the Office for Violence Against Women (OVW) the Yale University team will evaluate the implementation process and impact of the U.S. Department of Justice's Domestic Violence Homicide Prevention Demonstration Initiative. This evaluation seeks to draw critical findings and potential lessons from the combined experience of the sites including: 1) how the models work in different communities; 2) the barriers and facilitators to implementing the models; and 3) outcomes of the model delivery. The evaluation team will also disseminate the findings with the goal of informing replication.

DETAILED DESCRIPTION:
Process Evaluation: The process evaluation will assess: 1) the training and technical assistance provided to sites; 2) the implementation of the models in the communities; and 3) characteristics of the service delivery systems.

Technical Assistance Providers will document the training and technical assistance (TTA) they provide to the sites.

Sites will be asked to identify key stakeholders to participate in interviews before the implementation begins and then two additional times during the demonstration phase. Key informant interviews will assess: recipient's perception of the training and technical assistance; model fidelity; model implementation (including model penetration, barriers and facilitators to implementation); and, perceptions of model impact. In addition to key informant interviews administrative data will be gathered to assess aspects of model implementation and systematic observations of law enforcement initiated screens will be conducted by a member of the evaluation team who will join patrol officers for "ride-alongs".

Impact Evaluation: The impact evaluation will assess changes in: 1) collaboration among service sectors; 2) supervision and sanctions for offenders; 3) recidivism and re-victimization; 4) victim reported feelings of safety; 5) utilization of resources; and 6) nature of safety planning.

System Collaboration will be assessed through a web-based survey completed at three time points by key stakeholders representing all potential partners in the community. Social network analysis will provide a visual depiction of how the network changes over time.

Victim Interviews will be conducted to determine the impact of involvement in the model program on their safety and wellbeing. Victims will be interviewed at three time points and will be asked about: prior and recent contact with law enforcement, domestic violence service providers or other providers; awareness of resources to address IPV; their safety and fear of their partner; coping strategies utilized; social support; financial resources; willingness to utilize criminal justice system and domestic violence service providers; both their and offenders behavior, beliefs and attitudes; self-reported mental health and substance abuse; their report of offenders substance abuse; and demographic information.

Administrative Data will be utilized to examine the breadth of the model implementation; the impact of the model programs on criminal justice processes; and whether there is a connection between the extent of post-risk assessment sanctions and services and the pattern of newly recorded incidents between the victim and offender. The evaluation will compare processing and outcomes across cases that are in many ways similar except that some cases were determined to be high risk and a risk assessment was completed and others where a risk assessment was not conducted. To facilitate these comparisons, the evaluation team will build a comprehensive database that will depict the "life-history" of each victim and offender dyad.

ELIGIBILITY:
The demonstration sites are:

California North Carolina Ohio Illinois Michigan Tennessee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all domestic violence offenders and victims within the six communities.
Sampling Method: Non-Probability Sample
Enrollment: 666 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Decreased frequency of re-assault | up to 3 years
  Decrease in harassment, assault, injury, homicide/mortality

SECONDARY OUTCOMES:
Increased collaboration between network partners | up to 3 years
  Increased information sharing, case planning, coordinated response
Increased awareness of and utilization of resources for victims | Up to 3 years
  Increased awareness of and utilization of community resources
Increased safety planning | Up to 3 years
  Increased safety planning at the time of police intervention
Increased victim reported safety | Up to 3 years
  Victim reported changes in perceptions of safety
Increased sanctions for offender | Up to 3 years
  Sanctions such as pre-trial containment, cases to trial, adjudications, containment post-adjudication

CONTACTS AND LOCATIONS:
Overall Officials: Joy S Kaufman, PhD, Principal Investigator — Yale University; Christopher Maxwell, PhD, Study Director — Michigan State University; Tami Sullivan, PhD, Study Director — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be archived with the National Institute of Justice
Supporting Information: Study Protocol, SAP
Time Frame: before December 31, 2020
Access Criteria: To be determined